CLINICAL TRIAL: NCT00101270
Title: A Phase I Study of Oxaliplatin (NSC# 266046, IND #57004) and Irinotecan in Pediatric Patients With Refractory Solid Tumors and Lymphomas
Brief Title: Oxaliplatin and Irinotecan in Treating Young Patients With Refractory Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01819; ADVL0415; CDR0000401518; COG-ADVL0415; U01CA097452 (NIH)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Childhood Burkitt Lymphoma; Childhood Central Nervous System Germ Cell Tumor; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Liver Cancer; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Medulloblastoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway Glioma; Recurrent Colon Cancer; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Melanoma; Recurrent Nasopharyngeal Cancer; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Recurrent/Refractory Childhood Hodgkin Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Astrocytoma; Familial ependymoma; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Optic Nerve Glioma; Colonic Neoplasms; Neuroectodermal Tumors, Primitive, Peripheral; Melanoma; Nasopharyngeal Neoplasms; Neuroblastoma; Osteosarcoma; Wilms Tumor; Recurrence | interventions — Irinotecan; Oxaliplatin

ARMS (1):
- Treatment (irinotecan hydrochloride, oxaliplatin) (Experimental): Patients receive oxaliplatin IV over 2 hours on days 1 and 8 and irinotecan IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: oxaliplatin

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP

SUMMARY:
This phase I trial is studying the side effects and best dose of oxaliplatin when given together with irinotecan in treating young patients with refractory solid tumors or lymphomas. Drugs used in chemotherapy, such as oxaliplatin and irinotecan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Oxaliplatin may help irinotecan kill more cancer cells by making cancer cells more sensitive to the drug. Giving oxaliplatin together with irinotecan may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of oxaliplatin when administered with irinotecan in pediatric patients with refractory solid tumors or lymphomas.

II. Determine the toxic effects of this regimen in these patients. III. Determine the pharmacokinetics of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine, preliminarily, the antitumor activity of this regimen in these patients.

II. Correlate UGT and BCRP genotype with the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of oxaliplatin.

Patients receive oxaliplatin IV over 2 hours on days 1 and 8 and irinotecan IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed refractory malignant solid tumor or lymphoma

  * Intrinsic brain stem tumors and optic pathway tumors do not require histologic verification
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life exists
* Measurable or evaluable disease

  * Evaluable disease is defined as a tumor that cannot be measured using a ruler or calipers, but can be assessed to determine disease progression or complete response, such as any of the following:

    * Positive lesions on metaiodobenzylguanidine (MIBG) or bone scan
    * Metastatic bone marrow disease
    * Elevated tumor markers
    * Presence of a malignant pleural effusion
* No leukemia
* Performance status - Karnofsky 50-100% (for patients > 10 years of age)
* Performance status - Lansky 50-100% (for patients ≤ 10 years of age)
* Not specified
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min
* Creatinine based on age as follows:

  * No greater than 0.8 mg/dL (for patients age 5 and under)
  * No greater than 1.0 mg/dL (for patients age 6 to 10)
  * No greater than 1.2 mg/dL (for patients age 11 to 15)
  * No greater than 1.5 mg/dL (for patients age 16 and over)
* No arrhythmia on EKG
* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry > 94% on room air and no evidence of pulmonary fibrosis by chest radiograph* or CT scan
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight ≥ 10 kg
* Neurologic deficits relatively stable for ≥ 1 week before study entry (patients with CNS tumors only)
* No electrolyte (e.g., sodium, potassium, bicarbonate, calcium, magnesium, and phosphate) abnormality ≥ grade 2 (electrolyte supplementation allowed)
* No uncontrolled infection
* No history of life-threatening allergy to camptothecin derivatives or platinum agents
* No sensory or motor peripheral neuropathy ≥ grade 2
* No elevation of amylase or lipase ≥ grade 2
* Able to tolerate enteral medications (e.g., cefixime, cefpodoxime, or loperamide)
* Recovered from all prior immunotherapy
* At least 7 days since prior hematopoietic growth factors
* At least 7 days since prior antineoplastic biologic therapy
* Prior stem cell transplantation or rescue without total-body irradiation (TBI) allowed provided ≥ 3 months have elapsed and there is no evidence of active graft-versus-host disease
* No concurrent immunotherapy
* No concurrent biologic therapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered
* No prior oxaliplatin
* No other concurrent chemotherapy
* Concurrent steroids allowed provided dose has been stable for ≥ 7 days before study entry
* See Biologic therapy
* Recovered from all prior radiotherapy
* At least 2 weeks since prior local palliative small port radiotherapy
* At least 6 months since prior TBI
* At least 6 months since prior craniospinal, whole spinal, or whole lung/abdominal radiotherapy
* At least 6 months since prior radiotherapy to ≥ 50 % of the pelvis
* At least 6 weeks since other prior substantial radiotherapy to the bone marrow
* No concurrent radiotherapy
* No other concurrent investigational drugs
* No other concurrent anticancer therapy
* No concurrent cephalosporin antibiotics
* No concurrent use of any of the following:

  * Phenytoin
  * Carbamazepine
  * Oxcarbazepine
  * Barbiturates
  * Rifampin
  * Phenobarbital
  * Azole antifungal agents
  * Aprepitant
  * Hypericum perforatum (St. John's wort)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
MTD of oxaliplatin, defined as the maximum dose at which fewer than one-third of patients experience DLT | 21 days
  Graded using the NCI CTCAE version 3.0.

SECONDARY OUTCOMES:
Overall response assessed using RECIST criteria | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa McGregor, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States